CLINICAL TRIAL: NCT05086822
Title: A Phase Ia Study on Tolerability and Pharmacokinetics of Irinotecan Hydrochloride Liposome Alone in Patients With Advanced Solid Tumors
Brief Title: A Study of Irinotecan Hydrochloride Liposome in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YLTKL-Ia-1
Record Dates: First submitted 2021-09-29; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — irinotecan sucrosofate

STUDY DESIGN:
Intervention Model Description: A dose-escalation（3+3 design） and expansion study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group A (Experimental): Treatment group : Irinotecan liposome
  Interventions: Drug: Irinotecan liposome

INTERVENTIONS:
Drug: Irinotecan liposome — Irinotecan liposome

SUMMARY:
This is an open label, dose-escalation and expansion, single centre, phase Ia study . In this study, the tolerability, safety, pharmacokinetics and efficacy of irinotecan hydrochloride liposome injection were studied in patients with advanced solid tumors, to determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of irinotecan hydrochloride liposome.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid tumors documented as advanced or metastatic disease;
2. Subjects must be considered relapsed or refractory to standard therapies, have been intolerant to standard therapies, or have refused standard therapy;
3. ECOG: 0-1;
4. Adequate organ and bone marrow function;
5. sign an informed consent.

Exclusion Criteria:

1. Patients with brain malignant tumor, lymphoma or other malignant hematologic diseases;
2. Active CNS metastasis;
3. Clinically significant GI disorders;
4. Significant cardiovascular disease;
5. Active infection or uncontrolled fever;
6. Pregnant or breast feeding patients;
7. Allergic to a drug ingredient or component;
8. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Adverse Event (AE) | Assessed from study inclusion to 30 days after last dose
  Assessed by CTCAE 4.03
Dose Limiting Toxicities (DLT) | DLTs will be evaluated during 21-day period following the first dose of study treatment
  Dose limiting toxicities for patients in the treatment
Maximal tolerated dose (MTD) | after the last patient in each cohort up to 12 months
  Maximum tolerated dose for patients in the treatment

SECONDARY OUTCOMES:
Objective Response Rate | maximum time on study 12 months
  Objective response rate was based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
Progression Free Survival | The maximum time in follow up was 12 months
  Progression-free survival was defined as the time from the date of randomization to the date of disease progression, or death (any cause) on or prior to the clinical cutoff date, whichever occurs first.
Time to reach maximum plasma concentration (Tmax) | up to 120 hours after the first dose
  Tmax of total irinotecan, free irinotecan and SN-38
Maximum observed plasma concentration (Cmax) | up to 120 hours after the first dose
  Cmax of total irinotecan, free irinotecan and SN-38
Area under the plasma concentration versus time curve from time zero to time of last observed concentration (AUC0-t) | up to 120 hours after the first dose
  AUC0-t of total irinotecan, free irinotecan and SN-38
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-inf) | up to 120 hours after the first dose
  AUC0-inf of total irinotecan, free irinotecan and SN-38
Elimination half-life (T1/2) | up to 120 hours after the first dose
  T1/2 of total irinotecan, free irinotecan and SN-38
Clearance of drug from plasma (CL) | up to 120 hours after the first dose
  CL of total irinotecan
Volume of distribution (Vss) | up to 120 hours after the first dose
  Vss of total irinotecan

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided